CLINICAL TRIAL: NCT01882816
Title: A Phase II Study of Intensity-Modulated Radiation Therapy (IMRT) in the Treatment of Non-Anaplastic Non-Medullary Thyroid Cancer
Brief Title: Intensity-Modulated Radiation Therapy (IMRT) in the Treatment of Non-Anaplastic Non-Medullary Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-070
Record Dates: First submitted 2013-06-13; First posted 2013-06-20 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2021-11

CONDITIONS: Thyroid Cancer
Keywords: non-anaplastic; non-medullary; radiation; IMRT; Doxorubicin; 13-070
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Diffusion Magnetic Resonance Imaging; Doxorubicin

ARMS (1):
- IMRT and doxorubicin (Experimental): All patients will undergo radiation treatments using IMRT with concurrent low-dose radiosensitizing doxorubicin at 10 mg/m2 will be administered.
  Interventions: Radiation: IMRT; Device: DWI MRI; Drug: Doxorubicin; Other: Modified Barium Swallow Impairment Profile (MBSImP)

INTERVENTIONS:
Radiation: IMRT — Patients will receive intensity-modulated radiation therapy (IMRT) in once-daily fractions (Monday through Friday, excluding holidays). A total dose of 70Gy is planned. Patients will be seen weekly during radiation as per standard procedure at MSKCC
Device: DWI MRI — The DW and multiparametric MRI will be recommended for 3 months, 6 months, and then every 6 months (all +/- 4 weeks) until 2 years post-RT unless contraindicated for main campus patients only. This schedule may be altered, as clinically indicated.
Drug: Doxorubicin — Low dose radiosensitizing doxorubicin at 10 mg/m2 will be administered weekly.
Other: Modified Barium Swallow Impairment Profile (MBSImP) — The MBSImP is a standardized tool which assesses swallowing impairment as it relates to oral, pharyngeal, and esophageal impairments.

SUMMARY:
The purpose of this Phase 2 study is to find out what effect, good and/or bad, external beam radiation therapy, has on the patient and their thyroid cancer where surgery is not an option or where despite surgery, the disease is still present.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of non-anaplastic non-medullary thyroid cancer that is either grossly recurrent after surgery or unresectable with or without metastatic disease.
* Age ≥18 years
* Karnofsky performance status ≥70%
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months after treatment.
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Women who are pregnant or lactating
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- [Derived] Romesser PB, Sherman EJ, Whiting K, Ho ML, Shaha AR, Sabra MM, Riaz N, Waldenberg TE, Sabol CR, Ganly I, McBride SM, Fagin JA, Zhang Z, Tuttle RM, Wong RJ, Lee NY. Intensity-modulated radiation therapy and doxorubicin in thyroid cancer: A prospective phase 2 trial. Cancer. 2021 Nov 15;127(22):4161-4170. doi: 10.1002/cncr.33804. Epub 2021 Jul 22. PMID 34293201
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMRT and Doxorubicin
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IMRT and Doxorubicin
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 45.6 [42.0 to 51.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local-regional Progression-free Survival
Description: 2-year cumulative incidence of locoregional progression/failure with death as a competing risk will be defined as infield progression if included in the RT field and meets one of the following criteria: 25% increase in tumor volume, new lesions, and/or 25% increase in metabolic tumor volume or total lesion glycolysis.
Time Frame: 2 years
Measure: Number; unit: percentage of all participants
Arm/Group | IMRT and Doxorubicin
Number analyzed (Participants) | 27
percentage of all participants | 15.2

2. Secondary Outcome: Overall Survival
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants alive
Arm/Group | IMRT and Doxorubicin
Number analyzed (Participants) | 27
percentage of participants alive | 77.3 [62.8 to 95.1]

3. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Treatment-related Toxicities
Description: During radiation, adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events-Version 4.0 Physician-reported acute grade 3 or higher treatment-related toxicities, regardless of attribution.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | IMRT and Doxorubicin
Number analyzed (Participants) | 27
percentage of participants | 33.4

4. Secondary Outcome: Rate of Late Dysphagia
Description: Grade 2 or higher late toxicity rate. During radiation, adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events-Version 4.0
Time Frame: 2 years
Measure: Number; unit: percent of pts experiencing dysphagia
Arm/Group | IMRT and Doxorubicin
Number analyzed (Participants) | 27
percent of pts experiencing dysphagia | 8.0

5. Secondary Outcome: Rate of Late Xerostomia/Dry Mouth
Description: Rate of late xerostomia/dry mouth. During radiation, adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events-Version 4.0
Time Frame: 2 years
Measure: Number; unit: percent of pts experiencing dry mouth
Arm/Group | IMRT and Doxorubicin
Number analyzed (Participants) | 27
percent of pts experiencing dry mouth | 4.0

6. Secondary Outcome: Number of Participants With Significant Functional Difference in Dysphagia at 12 Months Compared to Baseline
Description: Comparison of significant functional differences 12 months after treatment assessed using standard Modified Barium Swallow Study
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | IMRT and Doxorubicin
Number analyzed (Participants) | 27
Participants
  Participants with significant functional difference as compared to baseline | 0
  Participants without significant functional difference as compared to baseline | 27

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | IMRT and Doxorubicin
All-Cause Mortality (participants affected / at risk) | 11/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 22/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT and Doxorubicin (N=27)
Stoma site infection (Infections and infestations) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT and Doxorubicin (N=27)
Anemia (Blood and lymphatic system disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 3
Lymphocyte count decreased (Investigations) | 22
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 3
White blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT01882816/Prot_SAP_000.pdf